CLINICAL TRIAL: NCT02314923
Title: A Phase 1 Randomized, Multi-Center, Double-Blind, Placebo-Controlled, Dose-Response Study to Evaluate the Safety and Immunogenicity of the BPSC-1001 (VSVΔG-ZEBOV) Ebola Virus Vaccine Candidate in Healthy Adult Subjects
Brief Title: Placebo Controlled, Dose Response, Safety and Immunogenicity Study of Vesicular Stomatitis Virus (VSV) Ebola Vaccine in Healthy Adults (V920-004)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: BioProtection Systems Corporation (Industry); Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V920-004; NLG0507 (Other: NewLink Genetics Corp.); V920-004 (Other: Merck Protocol Number)
Record Dates: First submitted 2014-12-08; First posted 2014-12-11 (Estimated); Results first posted 2020-01-02 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Ebola Virus

STUDY DESIGN:
Intervention Model Description: The study comprised two separate cohorts. Cohort 1 consisted of the 4 lower V920 dose groups (3x10^3 pfu, 3x10^4 pfu, 3x10^5 pfu, and 3x10^6 pfu). Cohort 2 consisted of the 3 higher V920 dose groups (9x10^6 pfu, 2x10^7 pfu, 1x10^8 pfu) plus a bridging group that received vaccine at the highest dose evaluated in Cohort 1 (i.e. 3x10^6 pfu). Both Cohorts 1 and 2 had a placebo group.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (10):
- 3x10^3 pfu Vaccine Cohort 1 (Experimental): Participants will receive a 1-mL intramuscular injection of V920 3x10^3 pfu in the deltoid on Day 0.
  Interventions: Biological: V920 Vaccine
- 3x10^4 pfu Vaccine Cohort 1 (Experimental): Participants will receive a 1-mL intramuscular injection of V920 3x10^4 pfu in the deltoid on Day 0.
  Interventions: Biological: V920 Vaccine
- 3x10^5 pfu Vaccine Cohort 1 (Experimental): Participants will receive a 1-mL intramuscular injection of V920 3x10^5 pfu in the deltoid on Day 0.
  Interventions: Biological: V920 Vaccine
- 3x10^6 pfu Vaccine Cohort 1 (Experimental): Participants will receive a 1-mL intramuscular injection of V920 3x10^6 pfu in the deltoid on Day 0.
  Interventions: Biological: V920 Vaccine
- 9x10^6 pfu Vaccine Cohort 2 (Experimental): Participants will receive a 1-mL intramuscular injection of V920 9x10^6 pfu in the deltoid on Day 0.
  Interventions: Biological: V920 Vaccine
- 2x10^7 pfu Vaccine Cohort 2 (Experimental): Participants will receive a 1-mL intramuscular injection of V920 2x10^7 pfu in the deltoid on Day 0.
  Interventions: Biological: V920 Vaccine
- 1x10^8 pfu Vaccine Cohort 2 (Experimental): Participants will receive a 1-mL intramuscular injection of V920 1x10^8 pfu in the deltoid on Day 0.
  Interventions: Biological: V920 Vaccine
- Placebo Cohort 1 (Placebo Comparator): Participants will receive a 1-mL intramuscular injection of placebo in the deltoid on Day 0.
  Interventions: Other: Placebo
- 3x10^6 pfu Vaccine Cohort 2 (Experimental): Participants will receive a 1-mL intramuscular injection of V920 3x10^3 pfu in the deltoid on Day 0.
  Interventions: Biological: V920 Vaccine
- Placebo Cohort 2 (Placebo Comparator): Participants will receive a 1-mL intramuscular injection of placebo in the deltoid on Day 0.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: V920 Vaccine — Vesicular Stomatitis Virus (VSV)-based vaccine 1-mL injection containing 3x10^3, 3x10^4, 3x10^5, 3x10^6, 9x10^6, 2x10^7, or 1x10^8 pfu.
  Other Names: BPSC-1001
  Arms: 1x10^8 pfu Vaccine Cohort 2; 2x10^7 pfu Vaccine Cohort 2; 3x10^3 pfu Vaccine Cohort 1; 3x10^4 pfu Vaccine Cohort 1; 3x10^5 pfu Vaccine Cohort 1; 3x10^6 pfu Vaccine Cohort 1; 3x10^6 pfu Vaccine Cohort 2; 9x10^6 pfu Vaccine Cohort 2
Other: Placebo — 0.9% Saline
  Arms: Placebo Cohort 1; Placebo Cohort 2

SUMMARY:
Ebola virus has infected and killed people, mostly in Africa. In 2014, the Ebola virus has affected several thousand people. There is no approved effective way to treat or prevent Ebola. Researchers are trying to develop a vaccine for it. This is a study of the anti-Ebola vaccine BPSC-1001 to see if it is safe and to see how it affects people's immune system.

DETAILED DESCRIPTION:
Between 1994 and the present, there have been many Ebola viruses (EBOV) outbreaks affecting mostly central Africa. However, the 2014 West African outbreak significantly exceeds all previous outbreaks in geographic range, number of individuals affected and in disruption of typical activities of civil society.

This is a Phase 1 safety and tolerability study to evaluate a novel vaccine to Ebola using a live replicating vesicular stomatitis virus (VSV) replacing the gene encoding the G envelope glycoprotein with the gene encoding the envelope glycoprotein from the Zaire strain of Ebola (VSVΔG-ZEBOV also known as V920 and BPSC-1001).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male or non-pregnant, non-lactating adult female, ages 18 to 60 (inclusive) at the time of screening
2. Have provided written informed consent prior to screening procedures
3. Free of clinically significant health problems, as determined by pertinent medical history, physical examination and clinical judgment of the investigator.
4. Available, able, and willing to participate for all study visits and procedures.
5. Males and females who are willing to practice abstinence from sexual intercourse with the opposite sex, or willing to use effective methods of contraception, from at least 30 days prior to vaccination until study end.
6. Be willing to minimize blood and body fluid exposure of others for 7 days after vaccination by:

   1. Using effective barrier prophylaxis, such as latex condoms, during penetrative sexual intercourse
   2. Avoiding the sharing of needles, razors, or toothbrushes
   3. Avoiding open-mouth kissing
7. Resides in the geographic area of a clinical study site for 1 year after vaccination without risk of deployment outside the U.S.

Exclusion Criteria:

1. History of prior infection with a filovirus or prior participation in a filovirus vaccine trial
2. History of prior infection with VSV or receipt of a VSV vectored vaccine
3. Has been involved in the care in any capacity of a patient with Ebola virus infection within the previous 21 days
4. Is a healthcare worker who has direct contact with patients (nurse, physician, dentist, emergency medical technician, dental hygienist)
5. Has a house-hold contact (HHC) who is immunodeficient, on immunosuppressive medications, human immunodeficiency virus (HIV)-positive, pregnant, has an unstable medical condition
6. Has an HHC, or is a childcare worker who has direct contact with children, 5 years of age or younger
7. Direct hands-on job preparing food in the food industry
8. History of employment in an industry involved in contact with ruminant animals, veterinary sciences, or other potential exposure to VSV
9. History of employment or activity which involves potential contact with filoviruses
10. History of severe local or systemic reactions to any vaccination or a history of severe allergic reactions
11. Known allergy to the components of the BPSC1001 vaccine product
12. Receipt of investigational product up to 30 days prior to randomization or ongoing participation in another clinical trial
13. Receipt of licensed non-live vaccines within 14 days of planned study immunization (30 days for live vaccines)
14. Ability to observe possible local reactions at the eligible injections sites (deltoid region) is, in the opinion of the investigator, unacceptably obscured due to a physical condition or permanent body art
15. Acute or chronic, clinically significant psychiatric, hematologic, pulmonary, cardiovascular, or hepatic or renal functional abnormality as determined by the investigator based on medical history, physical examination, and/or laboratory screening test. This would include a known hemoglobinopathy or coagulation abnormality.
16. Any baseline laboratory screening test which in the opinion of the investigator, is considered clinically significant
17. Any serologic evidence of hepatitis B or C infection
18. Any confirmed or suspected immunosuppressive or immunodeficient condition, including HIV-1, HIV-2 infection, cytotoxic therapy in the previous 5 years, and/or diabetes
19. Any chronic or active neurologic disorder, including migraines, seizures, and epilepsy, excluding a single febrile seizure as a child
20. Have a known history of Guillain-Barré Syndrome
21. Have an active malignancy or history of metastatic or hematologic malignancy
22. Suspected or known alcohol and/or illicit drug abuse within the past 5 years
23. Moderate or severe illness and/or fever >100.4°F within 1 week prior to vaccination (can be rescheduled)
24. Pregnant or lactating female, or female who intends to become pregnant during the study period
25. Administration of IgGs and/or any blood products within the 120 days preceding study entry or planned administration during the study period
26. History of blood donation within 60 days of enrollment or plans to donate within the study period
27. Administration of chronic (defined as more than 14 days) immunosuppressants or other immune modifying drugs within 6 months of study entry

    1. For corticosteroids, this includes prednisone, or equivalent, greater than or equal to 0.5 mg/kg/day
    2. Intranasal, topical, and intra-articular steroids are allowed
28. Unwilling to allow storage and use of blood for future vaccine research

28. Research staff or the immediate family of research staff directly involved with the clinical study.

29. Unwilling to undergo diagnostic evaluation of joint signs and symptoms, which may include arthrocentesis if clinically indicated based on presence of effusion and if the procedure is acceptable to the subject at the time (Cohort 2 only) 30. Unwilling to undergo diagnostic evaluation of skin rash, to include punch biopsy if clinically indicated and if the procedure is acceptable to the subject at the time (Cohort 2 only) 31. Research staff or the immediate family of research staff directly involved in the clinical study 32. Any other significant finding that in the opinion of the investigator would increase the risk of the individual having an adverse outcome from participating in this study 33. Elective surgery or hospitalization planned during the period of study participation 34. Has traveled to an area where the World Health Organization has declared as an Ebola outbreak zone 35. History of chronic inflammatory disease (e.g., rheumatoid arthritis, psoriatic arthritis, reactive arthritis, ankylosing spondylitis, systemic lupus erythematosus, psoriasis, Crohn's disease, ulcerative colitis, and gout), symptomatic osteoarthritis, or any other autoimmune or autoinflammatory disorder

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 513 (Actual)
Dates: Start 2014-12-05 (Actual); Primary Completion 2016-06-23 (Actual); Study Completion 2016-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Heppner DG Jr, Kemp TL, Martin BK, Ramsey WJ, Nichols R, Dasen EJ, Link CJ, Das R, Xu ZJ, Sheldon EA, Nowak TA, Monath TP; V920-004 study team. Safety and immunogenicity of the rVSV∆G-ZEBOV-GP Ebola virus vaccine candidate in healthy adults: a phase 1b randomised, multicentre, double-blind, placebo-controlled, dose-response study. Lancet Infect Dis. 2017 Aug;17(8):854-866. doi: 10.1016/S1473-3099(17)30313-4. Epub 2017 Jun 9. PMID 28606591
- [Derived] Coller BG, Blue J, Das R, Dubey S, Finelli L, Gupta S, Helmond F, Grant-Klein RJ, Liu K, Simon J, Troth S, VanRheenen S, Waterbury J, Wivel A, Wolf J, Heppner DG, Kemp T, Nichols R, Monath TP. Clinical development of a recombinant Ebola vaccine in the midst of an unprecedented epidemic. Vaccine. 2017 Aug 16;35(35 Pt A):4465-4469. doi: 10.1016/j.vaccine.2017.05.097. Epub 2017 Jun 21. PMID 28647166

RESULTS

PARTICIPANT FLOW:
Groups:
- 3x10^3 Plaque-forming Units (Pfu) V920: Cohort 1: Participants received a single 1.0 mL intramuscular injection of V920 3x10^3 pfu in the deltoid on Day 0.
- 3x10^4 Pfu V920: Cohort 1: Participants received a single 1.0 mL intramuscular injection of V920 3x10^4 pfu in the deltoid on Day 0.
- 3x10^5 Pfu V920: Cohort 1: Participants received a single 1.0 mL intramuscular injection of V920 3x10^5 pfu in the deltoid on Day 0.
- 3x10^6 Pfu V920: Cohort 1: Participants received a 1.0 mL intramuscular injection of V920 3x10^6 pfu in the deltoid on Day 0.
- Placebo: Cohort 1; Placebo: Cohort 2: Participants received a single 1.0 mL intramuscular injection of placebo in the deltoid on Day 0.
- 3x10^6 Pfu V920: Cohort 2: Participants received a single 1.0 mL intramuscular injection of V920 3x10^6 pfu in the deltoid on Day 0
- 9x10^6 Pfu V920: Cohort 2: Participants received a 1.0 mL intramuscular injection of V920 9x10^6 pfu in the deltoid on Day 0.
- 2x10^7 Pfu V920: Cohort 2: Participants received a single 1.0 mL intramuscular injection of V920 2x10^7 pfu in the deltoid on Day 0.
- 1x10^8 Pfu V920: Cohort 2: Participants received a single 1.0 mL intramuscular injection of V920 1x10^8 pfu in the deltoid on Day 0.
Period: Overall Study
Arm/Group | 3x10^3 Plaque-forming Units (Pfu) V920: Cohort 1 | 3x10^4 Pfu V920: Cohort 1 | 3x10^5 Pfu V920: Cohort 1 | 3x10^6 Pfu V920: Cohort 1 | Placebo: Cohort 1 | 3x10^6 Pfu V920: Cohort 2 | 9x10^6 Pfu V920: Cohort 2 | 2x10^7 Pfu V920: Cohort 2 | 1x10^8 Pfu V920: Cohort 2 | Placebo: Cohort 2
Started | 64 | 64 | 64 | 64 | 74 | 20 | 48 | 47 | 48 | 20
Treated | 64 | 64 | 64 | 64 | 74 | 20 | 47 (One participant did not receive vaccination due to missing blood sample at randomization.) | 47 | 48 | 20
Completed | 61 | 60 | 62 | 63 | 73 | 19 | 43 | 42 | 46 | 20
Not Completed | 3 | 4 | 2 | 1 | 1 | 1 | 5 | 5 | 2 | 0
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 3 | 1 | 0 | 0 | 0 | 3 | 4 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Participant unavailable | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Screen failure | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Participant relocation | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were reported for treated participants. 1 participant in 9x10^6 pfu V920: Cohort 2 arm did not receive vaccine
Groups:
- 3x10^3 Pfu V920: Cohort 1: Participants received a single 1.0 mL intramuscular injection of V920 3x10^3 pfu in the deltoid on Day 0
- 3x10^4 Pfu V920: Cohort 1: Participants received a 1.0 mL intramuscular injection of V920 3x10^4 pfu in the deltoid on Day 0.
- 3x10^5 Pfu V920: Cohort 1: Participants received a 1.0 mL intramuscular injection of V920 3x10^5 pfu in the deltoid on Day 0.
- Placebo Cohort 1; Placebo: Cohort 2: Participants received a single 1.0 mL intramuscular injection of placebo in the deltoid on Day 0.
- 2x10^7 Pfu V920: Cohort 2: Participants received a 1.0 mL intramuscular injection of V920 2x10^7 pfu in the deltoid on Day 0.
- 1x10^8 Pfu V920: Cohort 2: Participants received a 1.0 mL intramuscular injection of V920 1x10^8 pfu in the deltoid on Day 0.
- Total: Total of all reporting groups
Arm/Group | 3x10^3 Pfu V920: Cohort 1 | 3x10^4 Pfu V920: Cohort 1 | 3x10^5 Pfu V920: Cohort 1 | 3x10^6 Pfu V920: Cohort 1 | Placebo Cohort 1 | 3x10^6 Pfu V920: Cohort 2 | 9x10^6 Pfu V920: Cohort 2 | 2x10^7 Pfu V920: Cohort 2 | 1x10^8 Pfu V920: Cohort 2 | Placebo: Cohort 2 | Total
Number analyzed (Participants) | 64 | 64 | 64 | 64 | 74 | 20 | 47 | 47 | 48 | 20 | 512
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 64 | 64 | 64 | 64 | 74 | 20 | 47 | 47 | 48 | 20 | 512
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 33 | 31 | 33 | 39 | 8 | 24 | 22 | 15 | 8 | 245
  Male | 32 | 31 | 33 | 31 | 35 | 12 | 23 | 25 | 33 | 12 | 267

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With One or More Solicited Injection-site Adverse Events by Severity
Description: An AE can be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study vaccine or protocol-specified procedure, whether or not considered related to the study vaccine or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the study vaccine or protocol-specified procedure is also an adverse event. Injection-site AEs prompted on the Vaccination Report Card (VRC) were erythema, pain, tenderness and swelling. AEs were assessed for severity by the investigator according to a toxicity grading scale based on the FDA Guidance for Industry: Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials. Grade 1=Mild; Grade 2=Moderate; Grade 3=Severe; Grade 4=Potentially life-threatening. The percentage of participants that experienced at least 1 solicited injection-site AE was summarized by grade.
Time Frame: Up to 14 days postvaccination
Population: All randomized participants who received study vaccination and had data available for the endpoint.
Measure: Number; unit: Percentage of Participants
Arm/Group | 3x10^3 Pfu V920: Cohort 1 | 3x10^4 Pfu V920: Cohort 1 | 3x10^5 Pfu V920: Cohort 1 | 3x10^6 Pfu V920: Cohort 1 | Placebo: Cohort 1 | 3x10^6 Pfu V920: Cohort 2 | 9x10^6 Pfu V920: Cohort 2 | 2x10^7 Pfu V920: Cohort 2 | 1x10^8 Pfu V920: Cohort 2 | Placebo: Cohort 2
Number analyzed (Participants) | 64 | 64 | 64 | 64 | 74 | 20 | 47 | 47 | 48 | 20
Percentage of Participants
  Grade 1 (Mild) | 17.2 | 21.9 | 29.7 | 45.3 | 10.8 | 30.0 | 61.7 | 63.8 | 47.9 | 5.0
  Grade 2 (Moderate) | 0 | 1.6 | 1.6 | 1.6 | 1.4 | 0 | 8.5 | 8.5 | 16.7 | 0
  Grade 3 (Severe) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 (Potentially life-threatening) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Percentage of Participants With One or More Solicited Systemic Adverse Events by Severity
Description: An AE can be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study vaccine or protocol-specified procedure, whether or not considered related to the study vaccine or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the study vaccine or protocol-specified procedure is also an adverse event. Systemic AEs included subjective and objective fever, shivering/chills, sweats, myalgia, arthralgia, joint swelling, joint tenderness, fatigue, headache, gastrointestinal symptoms (nausea, vomiting, abdominal pain, and diarrhea), mucosal lesion, and skin lesion (including any blisters). AEs were assessed for severity by the investigator as follows: Grade 1=Mild; Grade 2=Moderate; Grade 3=Severe; Grade 4=Potentially life-threatening. The percentage of participants that experienced at least one systemic AE was summarized by grade.
Time Frame: Up to 14 days postvaccination
Population: All randomized participants who received study vaccination and had data available for the endpoint.
Measure: Number; unit: Percentage of Participants
Arm/Group | 3x10^3 Pfu V920: Cohort 1 | 3x10^4 Pfu V920: Cohort 1 | 3x10^5 Pfu V920: Cohort 1 | 3x10^6 Pfu V920: Cohort 1 | Placebo: Cohort 1 | 3x10^6 Pfu V920: Cohort 2 | 9x10^6 Pfu V920: Cohort 2 | 2x10^7 Pfu V920: Cohort 2 | 1x10^8 Pfu V920: Cohort 2 | Placebo: Cohort 2
Number analyzed (Participants) | 64 | 64 | 64 | 64 | 74 | 20 | 47 | 47 | 48 | 20
Percentage of Participants
  Grade 1 (Mild) | 29.7 | 39.1 | 45.3 | 53.1 | 41.9 | 25.0 | 46.8 | 46.8 | 43.8 | 20.0
  Grade 2 (Moderate) | 10.9 | 4.7 | 10.9 | 14.1 | 4.1 | 25.0 | 19.1 | 23.4 | 27.1 | 5.0
  Grade 3 (Severe) | 0 | 0 | 3.1 | 1.6 | 0 | 0 | 2.1 | 4.3 | 4.2 | 0
  Grade 4 (Potentially life-threatening) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Percentage of Participants With One or More Unsolicited Vaccine-related Adverse Event by Severity
Description: An AE can be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study vaccine or protocol-specified procedure, whether or not considered related to the study vaccine or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the study vaccine or protocol-specified procedure is also an adverse event. Unsolicited vaccine-related AEs were those events not specifically listed as either an injection-site (local) or systemic in the VRC and were reported as at least possibly related to the study vaccine or placebo. The AEs were further assessed for severity by the investigator as follows: Grade 1=Mild; Grade 2=Moderate; Grade 3=Severe; Grade 4=Potentially life-threatening. The percentage of participants that experienced at least one unsolicited vaccine-related AE was summarized by grade..
Time Frame: Up to 56 days postvaccination
Population: All randomized participants who received study vaccination and had data available for the endpoint.
Measure: Number; unit: Percentage of Participants
Arm/Group | 3x10^3 Pfu V920: Cohort 1 | 3x10^4 Pfu V920: Cohort 1 | 3x10^5 Pfu V920: Cohort 1 | 3x10^6 Pfu V920: Cohort 1 | Placebo: Cohort 1 | 3x10^6 Pfu V920: Cohort 2 | 9x10^6 Pfu V920: Cohort 2 | 2x10^7 Pfu V920: Cohort 2 | 1x10^8 Pfu V920: Cohort 2 | Placebo: Cohort 2
Number analyzed (Participants) | 64 | 64 | 64 | 64 | 74 | 20 | 47 | 47 | 48 | 20
Percentage of Participants
  1 (Mild) | 7.8 | 14.1 | 7.8 | 9.4 | 6.8 | 15.0 | 14.9 | 17.0 | 14.6 | 10.0
  2 (Moderate) | 4.7 | 3.1 | 0 | 3.1 | 0 | 0 | 6.4 | 2.1 | 2.1 | 0
  3 (Severe) | 0 | 0 | 0 | 1.6 | 0 | 0 | 0 | 0 | 0 | 5.0
  4 (Potentially Life-threatening) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Percentage of Participants With One or More Serious Adverse Event (SAE) by Severity
Description: An adverse event is defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with study vaccine. An SAE is an AE that results in death, is life-threatening, results in a persistent or significant disability or incapacity, results in or prolongs an existing hospitalization, is a congenital anomaly or birth defect, or is another important medical event. SAEs were assessed for severity by the investigator as follows: Grade 1=Mild; Grade 2=Moderate; Grade 3=Severe; Grade 4=Potentially life-threatening; 5=Fatal. The percentage of participants that experienced at least 1 SAE was summarized by grade.
Time Frame: Up to 360 days postvaccination
Population: All randomized participants who received study vaccination and had data available for the endpoint.
Measure: Number; unit: Percentage of Participants
Arm/Group | 3x10^3 Pfu V920: Cohort 1 | 3x10^4 Pfu V920: Cohort 1 | 3x10^5 Pfu V920: Cohort 1 | 3x10^6 Pfu V920: Cohort 1 | Placebo: Cohort 1 | 3x10^6 Pfu V920: Cohort 2 | 9x10^6 Pfu V920: Cohort 2 | 2x10^7 Pfu V920: Cohort 2 | 1x10^8 Pfu V920: Cohort 2 | Placebo: Cohort 2
Number analyzed (Participants) | 64 | 64 | 64 | 64 | 74 | 20 | 47 | 47 | 48 | 20
Percentage of Participants
  1 (Mild) | 0 | 0 | 0 | 1.6 | 0 | 0 | 0 | 0 | 0 | 0
  2 (Moderate) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  3 (Severe) | 0 | 0 | 0 | 0 | 1.4 | 0 | 0 | 0 | 0 | 0
  4 (Potentially Life-threatening) | 0 | 0 | 1.6 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  5 (Fatal) | 0 | 0 | 0 | 1.6 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Geometric Mean Titers (GMTs) of Zaire Ebola Virus- (ZEBOV)-Specific Immunoglobulin-G (IgG) Antibody
Description: Blood was drawn on Day 28 to assess the GMTs of ZEBOV-specific IgG antibodies as determined by Enzyme-linked immunosorbent assay (ELISA).
Time Frame: 28 days postvaccination
Population: All participants who were vaccinated, had endpoint titer results on Days 0 (baseline) and 28 (relative Days 24-35), and who did not have any protocol violations that influenced interpretation of immunogenicity endpoints. A subset of 25 placebo recipients in Cohort 1 were prospectively identified for testing of immunogenicity endpoints.
Measure: Geometric Mean (Standard Deviation); unit: ELISA Units/mL
Arm/Group | 3x10^3 Pfu V920: Cohort 1 | 3x10^4 Pfu V920: Cohort 1 | 3x10^5 Pfu V920: Cohort 1 | 3x10^6 Pfu V920: Cohort 1 | Placebo: Cohort 1 | 3x10^6 Pfu V920: Cohort 2 | 9x10^6 Pfu V920: Cohort 2 | 2x10^7 Pfu V920: Cohort 2 | 1x10^8 Pfu V920: Cohort 2 | Placebo: Cohort 2
Number analyzed (Participants) | 64 | 61 | 64 | 63 | 25 | 20 | 45 | 46 | 45 | 20
ELISA Units/mL | 777.8 (5.06) | 767.8 (3.96) | 909.6 (3.26) | 1139.9 (3.25) | 30.3 (1.00) | 1518.9 (3.20) | 977.4 (3.01) | 1542.8 (3.10) | 1930.3 (2.22) | 35.9 (2.13)
Statistical Analysis 1: Comparison: 3x10^3 Pfu V920: Cohort 1 vs 3x10^4 Pfu V920: Cohort 1; Test type: Other; p = 0.951, ANOVA
Statistical Analysis 2: Comparison: 3x10^3 Pfu V920: Cohort 1 vs 3x10^5 Pfu V920: Cohort 1; Test type: Other; p = 0.458, ANOVA
Statistical Analysis 3: Comparison: 3x10^3 Pfu V920: Cohort 1 vs 3x10^6 Pfu V920: Cohort 1; Test type: Other; p = 0.071, ANOVA
Statistical Analysis 4: Comparison: 3x10^3 Pfu V920: Cohort 1 vs Placebo: Cohort 1; Test type: Other; p < 0.001, ANOVA
Statistical Analysis 5: Comparison: 3x10^3 Pfu V920: Cohort 1 vs 3x10^6 Pfu V920: Cohort 2; Test type: Other; p = 0.029, ANOVA
Statistical Analysis 6: Comparison: 3x10^3 Pfu V920: Cohort 1 vs 9x10^6 Pfu V920: Cohort 2; Test type: Other; p = 0.325, ANOVA
Statistical Analysis 7: Comparison: 3x10^3 Pfu V920: Cohort 1 vs 2x10^7 Pfu V920: Cohort 2; Test type: Other; p = 0.003, ANOVA
Statistical Analysis 8: Comparison: 3x10^3 Pfu V920: Cohort 1 vs 1x10^8 Pfu V920: Cohort 2; Test type: Other; p < 0.001, ANOVA
Statistical Analysis 9: Comparison: 3x10^4 Pfu V920: Cohort 1 vs 3x10^5 Pfu V920: Cohort 1; Test type: Other; p = 0.427, ANOVA
Statistical Analysis 10: Comparison: 3x10^4 Pfu V920: Cohort 1 vs 3x10^6 Pfu V920: Cohort 1; Test type: Other; p = 0.065, ANOVA
Statistical Analysis 11: Comparison: 3x10^4 Pfu V920: Cohort 1 vs Placebo: Cohort 1; Test type: Other; p < 0.001, ANOVA
Statistical Analysis 12: Comparison: 3x10^4 Pfu V920: Cohort 1 vs 3x10^6 Pfu V920: Cohort 2; Test type: Other; p = 0.027, ANOVA
Statistical Analysis 13: Comparison: 3x10^4 Pfu V920: Cohort 1 vs 9x10^6 Pfu V920: Cohort 2; Test type: Other; p = 0.303, ANOVA
Statistical Analysis 14: Comparison: 3x10^4 Pfu V920: Cohort 1 vs 2x10^7 Pfu V920: Cohort 2; Test type: Other; p = 0.003, ANOVA
Statistical Analysis 15: Comparison: 3x10^4 Pfu V920: Cohort 1 vs 1x10^8 Pfu V920: Cohort 2; Test type: Other; p < 0.001, ANOVA
Statistical Analysis 16: Comparison: 3x10^5 Pfu V920: Cohort 1 vs 3x10^6 Pfu V920: Cohort 1; Test type: Other; p = 0.286, ANOVA
Statistical Analysis 17: Comparison: 3x10^5 Pfu V920: Cohort 1 vs Placebo: Cohort 1; Test type: Other; p < 0.001, ANOVA
Statistical Analysis 18: Comparison: 3x10^5 Pfu V920: Cohort 1 vs 3x10^6 Pfu V920: Cohort 2; Test type: Other; p = 0.094, ANOVA
Statistical Analysis 19: Comparison: 3x10^5 Pfu V920: Cohort 1 vs 9x10^6 Pfu V920: Cohort 2; Test type: Other; p = 0.757, ANOVA
Statistical Analysis 20: Comparison: 3x10^5 Pfu V920: Cohort 1 vs 2x10^7 Pfu V920: Cohort 2; Test type: Other; p = 0.022, ANOVA
Statistical Analysis 21: Comparison: 3x10^5 Pfu V920: Cohort 1 vs 1x10^8 Pfu V920: Cohort 2; Test type: Other; p = 0.001, ANOVA
Statistical Analysis 22: Comparison: 3x10^6 Pfu V920: Cohort 1 vs Placebo: Cohort 1; Test type: Other; p < 0.001, ANOVA
Statistical Analysis 23: Comparison: 3x10^6 Pfu V920: Cohort 1 vs 3x10^6 Pfu V920: Cohort 2; Test type: Other; p = 0.348, ANOVA
Statistical Analysis 24: Comparison: 3x10^6 Pfu V920: Cohort 1 vs 9x10^6 Pfu V920: Cohort 2; Test type: Other; p = 0.508, ANOVA
Statistical Analysis 25: Comparison: 3x10^6 Pfu V920: Cohort 1 vs 2x10^7 Pfu V920: Cohort 2; Test type: Other; p = 0.191, ANOVA
Statistical Analysis 26: Comparison: 3x10^6 Pfu V920: Cohort 1 vs 1x10^8 Pfu V920: Cohort 2; Test type: Other; p = 0.024, ANOVA
Statistical Analysis 27: Comparison: 3x10^6 Pfu V920: Cohort 2 vs 9x10^6 Pfu V920: Cohort 2; Test type: Other; p = 0.169, ANOVA
Statistical Analysis 28: Comparison: 3x10^6 Pfu V920: Cohort 2 vs 2x10^7 Pfu V920: Cohort 2; Test type: Other; p = 0.961, ANOVA
Statistical Analysis 29: Comparison: 3x10^6 Pfu V920: Cohort 2 vs 1x10^8 Pfu V920: Cohort 2; Test type: Other; p = 0.454, ANOVA
Statistical Analysis 30: Comparison: 3x10^6 Pfu V920: Cohort 2 vs Placebo: Cohort 2; Test type: Other; p < 0.001, ANOVA
Statistical Analysis 31: Comparison: 9x10^6 Pfu V920: Cohort 2 vs 2x10^7 Pfu V920: Cohort 2; Test type: Other; p = 0.068, ANOVA
Statistical Analysis 32: Comparison: 9x10^6 Pfu V920: Cohort 2 vs 1x10^8 Pfu V920: Cohort 2; Test type: Other; p = 0.007, ANOVA
Statistical Analysis 33: Comparison: 9x10^6 Pfu V920: Cohort 2 vs Placebo: Cohort 2; Test type: Other; p < 0.001, ANOVA
Statistical Analysis 34: Comparison: 2x10^7 Pfu V920: Cohort 2 vs 1x10^8 Pfu V920: Cohort 2; Test type: Other; p = 0.370, ANOVA
Statistical Analysis 35: Comparison: 1x10^8 Pfu V920: Cohort 2 vs Placebo: Cohort 2; Test type: Other; p < 0.001, ANOVA

6. Secondary Outcome: Mean Copies of Vector Ribonucleic Acid (RNA) for Participants With a V920 Polymerase Chain Reaction (PCR) Result ≥ Lower Limit of Quantification (LLOQ)
Description: Participants had blood, assessed for evidence of V920 via polymerase chain reaction (PCR). Mean copies of RNA was reported for all participants who had reading ≥ the LLOQ (62.5 copies/mL)
Time Frame: Days 1, 2, 3, 4, 7, 14 and 28 post-vaccination
Population: as for outcome 5
Measure: Geometric Mean (Standard Deviation); unit: copies/mL
Arm/Group | 3x10^3 Pfu V920: Cohort 1 | 3x10^4 Pfu V920: Cohort 1 | 3x10^5 Pfu V920: Cohort 1 | 3x10^6 Pfu V920: Cohort 1 | Placebo: Cohort 1 | 3x10^6 Pfu V920: Cohort 2 | 9x10^6 Pfu V920: Cohort 2 | 2x10^7 Pfu V920: Cohort 2 | 1x10^8 Pfu V920: Cohort 2 | Placebo: Cohort 2
Number analyzed (Participants) | 64 | 61 | 64 | 63 | 25 | 20 | 45 | 46 | 45 | 20
copies/mL
  Day 1: number analyzed (Participants) | 0 | 0 | 0 | 5 | 0 | 1 | 10 | 9 | 27 | 0
  Day 1 |  |  |  | 118.04 (1.185) |  | 109.40 (NA) — SD could not be calculated due to low n | 144.72 (1.511) | 184.65 (1.893) | 304.45 (2.534) |
  Day 2: number analyzed (Participants) | 1 | 0 | 0 | 20 | 0 | 1 | 9 | 9 | 13 | 0
  Day 2 | 4107.00 (NA) — SD could not be calculated due to low n |  |  | 127.13 (1.511) |  | 109.40 (NA) — SD could not be calculated due to low n | 158.74 (1.901) | 172.24 (1.628) | 161.67 (1.644) |
  Day 3: number analyzed (Participants) | 1 | 1 | 0 | 3 | 0 | 0 | 0 | 1 | 3 | 0
  Day 3 | 12649.00 (NA) — SD could not be calculated due to low n | 109.40 (NA) — SD could not be calculated due to low n |  | 703.36 (25.106) |  |  |  | 109.40 (NA) — SD could not be calculated due to low n | 740.96 (8.199) |
  Day 4: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 4 | 23936.00 (NA) — SD could not be calculated due to low n | 109.40 (NA) — SD could not be calculated due to low n |  |  |  |  |  |  |  |
  Day 7: number analyzed (Participants) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 7 | 787.00 (NA) — SD could not be calculated due to low n |  | 160.00 (NA) — SD could not be calculated due to low n |  |  |  |  |  |  |
  Day 14: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Day 14 |  |  |  | 109.40 (NA) — SD could not be calculated due to low n |  |  |  |  |  |
  Day 28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Percentage of Participants With Seroconversion for ZEBOV-specific IgG
Description: Blood was drawn on Days 7, 14, 28, 56, 84 (Cohort 1 only), 180, and 360 days to assess the GMTs via ELISA. Seroconversion was defined as a post-vaccination titer ≥ 200 ELISA Units/mL that was also at least a 4-fold increase in titer compared to baseline.
Time Frame: 7, 14, 28, 56, 84 (Cohort 1 only), 180, and 360 days postvaccination
Population: as for outcome 5
Measure: Number; unit: Percentage of Participants
Arm/Group | 3x10^3 Pfu V920: Cohort 1 | 3x10^4 Pfu V920: Cohort 1 | 3x10^5 Pfu V920: Cohort 1 | 3x10^6 Pfu V920: Cohort 1 | Placebo: Cohort 1 | 3x10^6 Pfu V920: Cohort 2 | 9x10^6 Pfu V920: Cohort 2 | 2x10^7 Pfu V920: Cohort 2 | 1x10^8 Pfu V920: Cohort 2 | Placebo: Cohort 2
Number analyzed (Participants) | 64 | 61 | 64 | 63 | 25 | 20 | 45 | 46 | 45 | 20
Percentage of Participants
  Day 7: number analyzed (Participants) | 61 | 60 | 64 | 62 | 1 | 20 | 44 | 45 | 45 | 14
  Day 7 | 0 | 1.7 | 0 | 0 | 0 | 0 | 0 | 2.2 | 2.2 | 0
  Day 14: number analyzed (Participants) | 61 | 59 | 63 | 62 | 1 | 20 | 44 | 44 | 44 | 14
  Day 14 | 11.5 | 20.3 | 20.6 | 50.0 | 0 | 40.0 | 54.5 | 81.8 | 72.7 | 0
  Day 28 | 82.8 | 80.3 | 89.1 | 93.7 | 0 | 90.0 | 91.1 | 93.5 | 95.6 | 5.0
  Day 56: number analyzed (Participants) | 63 | 61 | 64 | 63 | 25 | 20 | 44 | 46 | 45 | 20
  Day 56 | 85.7 | 86.9 | 92.2 | 93.7 | 0 | 90.0 | 93.2 | 97.8 | 97.8 | 0
  Day 84: number analyzed (Participants) | 60 | 61 | 63 | 61 | 1 | 0 | 0 | 0 | 0 | 0
  Day 84 | 81.7 | 85.2 | 87.3 | 93.4 | 0 |  |  |  |  |
  Day 180: number analyzed (Participants) | 61 | 58 | 61 | 61 | 0 | 18 | 41 | 41 | 41 | 1
  Day 180 | 82.0 | 75.9 | 83.6 | 89.9 |  | 94.4 | 90.2 | 97.6 | 97.6 | 0
  Day 360: number analyzed (Participants) | 51 | 52 | 56 | 57 | 2 | 18 | 38 | 39 | 41 | 0
  Day 360 | 78.4 | 75.0 | 80.4 | 89.5 | 0 | 94.4 | 89.5 | 97.4 | 93.2 |
  Any time postvaccination | 89.1 | 90.2 | 93.8 | 96.8 | 0 | 100.0 | 97.8 | 97.8 | 97.8 | 5.0

8. Secondary Outcome: Percentage of Participants With Seroconversion for ZEBOV Neutralizing Antibodies
Description: Blood was drawn on Days 7, 14, 28, 56, 84 (Cohort 1 only), 180, and 360 days to assess the GMTs of Zaire ebolavirus neutralizing antibodies as determined plaque reduction neutralization titer (reciprocal of the dilution that resulted in a 60% decrease in plaques) (PRNT60).
Time Frame: 7, 14, 28, 56, 84 (Cohort 1 only), 180, and 360 days postvaccination
Population: as for outcome 5
Measure: Number; unit: Percentage of Participants
Arm/Group | 3x10^3 Pfu V920: Cohort 1 | 3x10^4 Pfu V920: Cohort 1 | 3x10^5 Pfu V920: Cohort 1 | 3x10^6 Pfu V920: Cohort 1 | Placebo: Cohort 1 | 3x10^6 Pfu V920: Cohort 2 | 9x10^6 Pfu V920: Cohort 2 | 2x10^7 Pfu V920: Cohort 2 | 1x10^8 Pfu V920: Cohort 2 | Placebo: Cohort 2
Number analyzed (Participants) | 64 | 61 | 64 | 63 | 25 | 20 | 45 | 46 | 45 | 20
Percentage of Participants
  Day 7: number analyzed (Participants) | 63 | 60 | 64 | 63 | 25 | 20 | 45 | 46 | 45 | 20
  Day 7 | 0 | 0 | 1.6 | 1.6 | 0 | 0 | 2.2 | 2.2 | 2.2 | 0
  Day 14: number analyzed (Participants) | 63 | 59 | 63 | 63 | 25 | 20 | 45 | 45 | 44 | 20
  Day 14 | 9.5 | 13.6 | 42.9 | 52.4 | 0 | 45.0 | 55.6 | 71.1 | 81.8 | 0
  Day 28: number analyzed (Participants) | 63 | 61 | 64 | 63 | 25 | 20 | 45 | 46 | 45 | 20
  Day 28 | 76.2 | 70.5 | 87.5 | 93.7 | 0 | 85.0 | 91.1 | 95.7 | 100.0 | 5.0
  Day 56: number analyzed (Participants) | 63 | 61 | 64 | 63 | 25 | 20 | 44 | 46 | 45 | 20
  Day 56 | 79.4 | 70.5 | 89.1 | 93.7 | 0 | 90.0 | 93.2 | 95.7 | 97.8 | 0
  Day 84 (Cohort 1 only): number analyzed (Participants) | 62 | 61 | 63 | 62 | 25 | 0 | 0 | 0 | 0 | 0
  Day 84 (Cohort 1 only) | 75.8 | 72.1 | 88.9 | 90.3 | 4.0 |  |  |  |  |
  Day 180: number analyzed (Participants) | 63 | 58 | 61 | 62 | 24 | 18 | 42 | 42 | 41 | 20
  Day 180 | 81.0 | 81.0 | 88.5 | 91.9 | 0 | 94.4 | 95.2 | 95.2 | 100.0 | 5.0
  Day 360: number analyzed (Participants) | 53 | 52 | 56 | 57 | 22 | 18 | 38 | 39 | 44 | 19
  Day 360 | 77.4 | 78.8 | 82.1 | 93.0 | 0 | 94.4 | 84.6 | 97.5 | 100.0 | 5.3
  Any time postvaccination | 89.1 | 88.5 | 96.9 | 98.4 | 4.0 | 100.0 | 97.8 | 100.0 | 100.0 | 10.0

9. Primary Outcome: Optimum Dose for General Use Prophylaxis With V920
Description: The optimum dose for general use prophylaxis with V920 was determined following the review of all immunogenicity and safety data.
Time Frame: Day 360
Population: All participants who received study vaccine
Measure: Number; unit: pfu
Groups:
- All Vaccinated Participants: All participants that received study vaccine.
Arm/Group | All Vaccinated Participants
Number analyzed (Participants) | 512
pfu | 20000000

ADVERSE EVENTS:
Time Frame: Up to 360 days
Description: All participants that received study vaccination (V920 dose or placebo).
Arm/Group | 3x10^3 Pfu V920: Cohort 1 | 3x10^4 Pfu V920: Cohort 1 | 3x10^5 Pfu V920: Cohort 1 | 3x10^6 Pfu V920: Cohort 1 | Placebo: Cohort 1 | 3x10^6 Pfu V920: Cohort 2 | 9x10^6 Pfu V920: Cohort 2 | 2x10^7 Pfu V920: Cohort 2 | 1x10^8 Pfu V920: Cohort 2 | Placebo: Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/64 | 0/64 | 1/64 | 0/74 | 0/20 | 0/47 | 0/47 | 0/48 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/64 | 1/64 | 2/64 | 1/74 | 0/20 | 0/47 | 0/47 | 0/48 | 0/20
Other Adverse Events (participants affected / at risk) | 30/64 | 38/64 | 44/64 | 52/64 | 43/74 | 14/20 | 43/47 | 41/47 | 41/48 | 9/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3x10^3 Pfu V920: Cohort 1 (N=64) | 3x10^4 Pfu V920: Cohort 1 (N=64) | 3x10^5 Pfu V920: Cohort 1 (N=64) | 3x10^6 Pfu V920: Cohort 1 (N=64) | Placebo: Cohort 1 (N=74) | 3x10^6 Pfu V920: Cohort 2 (N=20) | 9x10^6 Pfu V920: Cohort 2 (N=47) | 2x10^7 Pfu V920: Cohort 2 (N=47) | 1x10^8 Pfu V920: Cohort 2 (N=48) | Placebo: Cohort 2 (N=20)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3x10^3 Pfu V920: Cohort 1 (N=64) | 3x10^4 Pfu V920: Cohort 1 (N=64) | 3x10^5 Pfu V920: Cohort 1 (N=64) | 3x10^6 Pfu V920: Cohort 1 (N=64) | Placebo: Cohort 1 (N=74) | 3x10^6 Pfu V920: Cohort 2 (N=20) | 9x10^6 Pfu V920: Cohort 2 (N=47) | 2x10^7 Pfu V920: Cohort 2 (N=47) | 1x10^8 Pfu V920: Cohort 2 (N=48) | Placebo: Cohort 2 (N=20)
Abdominal pain (Gastrointestinal disorders) | 7 (9) | 3 (3) | 6 (7) | 2 (2) | 4 (5) | 0 (0) | 4 (4) | 3 (3) | 5 (5) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 6 (13) | 2 (3) | 6 (7) | 6 (7) | 8 (9) | 2 (2) | 7 (8) | 6 (7) | 11 (13) | 1 (1)
Nausea (Gastrointestinal disorders) | 9 (9) | 6 (7) | 13 (14) | 11 (13) | 12 (14) | 4 (4) | 4 (4) | 5 (7) | 6 (6) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (5) | 2 (2) | 4 (4) | 5 (5) | 4 (5) | 1 (1) | 1 (1) | 1 (1) | 3 (4) | 0 (0)
Chills (General disorders) | 6 (6) | 3 (3) | 7 (8) | 21 (22) | 6 (6) | 3 (3) | 16 (18) | 13 (14) | 15 (17) | 1 (1)
Fatigue (General disorders) | 12 (13) | 13 (16) | 14 (17) | 21 (24) | 14 (16) | 6 (6) | 17 (22) | 18 (25) | 22 (25) | 4 (6)
Pyrexia (General disorders) | 3 (3) | 4 (6) | 6 (6) | 16 (19) | 3 (3) | 6 (8) | 14 (18) | 18 (24) | 15 (20) | 0 (0)
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
Tenderness (General disorders) | 10 (10) | 12 (14) | 16 (17) | 26 (27) | 7 (7) | 4 (4) | 28 (29) | 28 (28) | 24 (24) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 6 (6) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 3 (3)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 2 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (18) | 11 (23) | 15 (23) | 11 (24) | 9 (13) | 4 (6) | 10 (22) | 11 (30) | 7 (21) | 2 (10)
Joint swelling (Musculoskeletal and connective tissue disorders) | 3 (5) | 2 (4) | 2 (2) | 3 (5) | 0 (0) | 1 (1) | 3 (3) | 4 (7) | 0 (0) | 1 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 12 (15) | 13 (16) | 15 (16) | 14 (15) | 10 (11) | 8 (12) | 19 (22) | 16 (18) | 16 (18) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 7 (7) | 12 (12) | 20 (20) | 6 (6) | 4 (4) | 28 (30) | 27 (28) | 25 (25) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 15 (24) | 19 (23) | 20 (27) | 32 (41) | 23 (33) | 7 (12) | 23 (32) | 22 (30) | 21 (28) | 3 (11)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 6 (7) | 3 (3) | 5 (5) | 5 (5) | 3 (5) | 4 (4) | 6 (7) | 11 (12) | 13 (15) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 3 (5) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data may be published in the open medical literature with the identity of the subjects protected. Anyone desiring to publish or present data obtained during the conduct of the study will conform to the Sponsor's policies and then forward the publication for review to the Sponsor prior to submission.